CLINICAL TRIAL: NCT04970082
Title: A Randomized Crossover Study to Evaluate and Compare the Reproducibility and Tolerability of Direct Wire Pacing for Measuring Fractional Flow Reserve Versus Standard Method in Subjects With FFR Indications
Brief Title: A Study to Evaluate Direct Wire Pacing (DWP) for Measuring Fractional Flow Reserve (FFR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Recherche Cardio Vasculaire Alpes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021-A00947-34
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Stenosis; Fractional Flow Reserve
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFR followed by FFR-DWP (investigation) (Experimental): The FFR measurement is performed with the standard method first followed by the FFR measurement with the DWP method.
  Interventions: Diagnostic Test: FFR DWP; Diagnostic Test: FFR
- FFR-DWP (investigation) followed by FFR (Experimental): The FFR measurement is performed with the DWP method first followed by the FFR measurement with the standard method.
  Interventions: Diagnostic Test: FFR DWP; Diagnostic Test: FFR

INTERVENTIONS:
Diagnostic Test: FFR DWP — FFR will be measured twice in the same lesion : One with the standard method and the other with the DWP method.
Diagnostic Test: FFR — FFR will be measured twice in the same lesion : One with the standard method and the other with the DWP method.

SUMMARY:
This is a randomized, non-inferiority, crossover investigation comparing the Direct Wire Pacing (DWP) versus standard method to measure Fractional Flow Reserve (FFR) in subjects with FFR indications.

All subjects requiring on a clinical basis a pressure wire assessment of coronary artery stenosis(es) will be eligible to take part in the study.

DETAILED DESCRIPTION:
Pressure wire-based Fractional Flow Reserve (FFR) has become the reference standard index of haemodynamic significance to guide revascularisation of intermediate coronary artery lesions.

The FFR measurement determines the ratio of the maximum blood flow that can be achieved in a diseased or narrowed coronary artery to the maximum blood flow in a normal coronary artery. This ratio represents the potential decrease in distal coronary flow relative to coronary stenosis.

FFR is easily measured during routine coronary angiography using a pressure wire to calculate the ratio of coronary pressure distal to a stenosis or diseased segment to aortic pressure under conditions of maximum myocardial hyperemia. An FFR of 1.0 is widely accepted as normal. An FFR of less than 0.80 is generally considered to be associated with coronary ischemia and widely accepted in favor of revascularization rather than conservative management.

The current standard method of measuring FFR is to insert a pressure wire into the coronary artery while the hyperaemic agent, usually adenosine, is delivered by intracoronary bolus or continuous intravenous injection.

Administration of adenosine may cause bradycardia and thus cause patient vagal discomfort. Direct Wire Pacing (DWP) can potentially overcome the drawbacks of the standard method when measuring FFR. Indeed, DWP allows to transmit an electrical current from the external pacemaker to the heart thanks to metallic FFR guidewire already used, and thus prevent bradycardia.

In addition, there are some absolute contraindications to the use of Adenosine such as 2nd or 3rd degree atrioventricular block, untreated sinus dysfunction or long QT syndrome ...DWP could allow this highly recommended diagnostic tool (1A) to be used in this patient population.

The investigators would therefore like to determine if the measurement of FFR by DWP would be non-inferior to the standard method to obtain precise FFR values and maximize patient's comfort.

ELIGIBILITY:
Eligible patient for coronary angiography.

Inclusion Criteria:

The patients included in the study must meet the following inclusion criteria :

* Patients ≥ 18 years old
* Patients with FFR indications
* Has given consent to undergo diagnostic coronary procedure
* Patients able to understand and provide informed consent
* Patients with Social Security coverage

Prior to randomisation: Angiography demonstrates at least one coronary stenosis in an artery, requiring FFR measurement for physiological assessment.

Exclusion Criteria:

The patients included in the study should not meet the following inclusion criteria :

* Contraindications to use sensitivity to Adenosine or any of its excipients
* Technically inaccessible stenosis(es)
* Pregnant or breastfeeding woman
* Patients under judicial protection, tutorship or curatorship
* Patient participating in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Reproducibility of the FFR measurement | Intraoperative
  Evaluated by the number of patients with comparable FFR ratio recording. The FFR ratio should remain constant (+/-0.02) between the two modes of measuring FFR.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Intraoperative
  Assessed by the number of participants with adverse events during the procedure.
Tolerance | Intraoperative
  Assessed by asking patients during each FFR to grade verbally any symptoms of chest discomfort.
correlation between a disproportionately high FFR value and la presence of a (partially) infarcted territory | Intraoperative
  The correlation between a disproportionately high FFR value in presence of a (partially)infarcted territory will be assessed by the comparison the obtained FFR value, the degree of angiographic stenosis measured and the obtained stimulation threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Faurie, Principal Investigator
Locations (1):
- Groupe Hospitalier Mutualiste de Grenoble, Grenoble, France